CLINICAL TRIAL: NCT00784992
Title: A Randomised Controlled Trial to Compare Success and Complication Rates in Endonasal Dacryocystorhinostomy Surgery With and Without Silicone Tubes
Brief Title: A Comparison of Endonasal Dacryocystorhinostomy With and Without Silicone Tubes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H08-02025
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Nasolacrimal Duct Obstruction
Keywords: NLDO; DCR; silicone tubes; stent
MeSH Terms: conditions — Lacrimal Duct Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Endonasal DCR with silicone tubes (this is the control group since it is the standard procedure / gold standard, although the evidence base for the use of tubes is lacking, hence the need for this trial)
- 2 (Active Comparator): Endonasal DCR without silicone tubes (this is the 'intervention' arm)
  Interventions: Procedure: Endonasal dacryocystorhinostomy

INTERVENTIONS:
Procedure: Endonasal dacryocystorhinostomy — The standard dacryocystorhinostomy operation performed in this centre uses silicone tubes to stent open the newly created ostium between the lacrimal sac and the nasal cavity. However many surgeons in other departments / countries around the world perform the surgery without tubes. No large well-conducted RCT has been published comparing success rates / complication rates for the two techniques. For this study the control group is the arm which receives tubes (our standard procedure) and the 'interventional' group is the arm not receiving tubes.
  Details of the operative technique for endonasal DCR with tubes can be found in the following reference: Dolman PJ. Comparison of external dacryocystorhinostomy with nonlaser endonasal dacryocystorhinostomy. Ophthalmology. 2003 Jan;110(1):78-84. The group that will not receive tubes will undergo the same procedure except that the insertion of tubes will be omitted.
  Arms: 2

SUMMARY:
Aim of study is to investigate whether the use of silicone tubes in endonasal DCR surgery increases the success rate and / or complication rate compared to surgery without tubes.

DETAILED DESCRIPTION:
Dacryocystorhinostomy (DCR) is the treatment of choice for epiphora due to nasolacrimal duct obstruction. A passage is created between the lacrimal sac and nasal cavity by removing the layers of bone and mucosa between them. It can be performed via an external (transcutaneous) or endonasal route with equivalent success rates.[1] In order to prevent restenosis of the ostium, silicone tubes are often used to maintain the patency of the newly-created fistula. The tubes are removed between 6 weeks and 3 months post-operatively.

Problems associated with tubes include granuloma formation with secondary infection or adhesions, canalicular lacerations, allergic reaction to the silastic, and discomfort.

There are a number of reports of DCR surgery without tubes which demonstrate an equivalent success rate compared with surgery using tubes; however, these studies have been non-randomised, retrospective reviews.[2-6] The only prospective, randomised controlled study[7] had only 42 participants and did not state at which point during the surgery the randomisation was revealed; unless the allocation occurs after the ostium has been completed there is the risk of bias since the surgeon may (consciously or inadvertently) create a larger ostium in cases where no tubes are to be used.

The purpose of this study is to perform a prospective, randomised controlled study to assess whether the use of tubes affect the long-term success of DCR.

Hypothesis Silicone tubing does not improve success rate of endonasal DCR surgery.

Justification There is a dearth of evidence in the literature from well-conducted studies on the merits of tubes versus no tubes in DCR surgery. Since there are several potential problems with tubes outlined above, and since performing surgery with tubes adds to the cost and duration of surgery, it would benefit patients and healthcare providers to know whether they increase DCR success rate.

The standard surgical technique for endonasal DCR has been described by the principle investigator.[1] The identical procedure would be performed in both groups with the exception that half the patients would have tubes inserted, and half would not.

Objectives To assess functional and anatomical success rates of endonasal DCR surgery with and without silicone tubes.

Research Method Prospective, randomised, controlled, interventional trial.

Statistical analysis The primary end point will be functional success, determined by patient-reported symptoms. This will be assessed a minimum of six months post-operatively. In patients with tubes these will be removed at 3 months post-operatively.

The operation will be considered successful if the patient is free of symptoms of a watering eye. It will be considered partially successful if the patient has noticeable improvement but still may experience tearing under certain situations. The operation will be deemed a failure if the patient continues to have symptoms that are no better or worse than pre-operatively.

The secondary end point will be anatomical success, as measured by patency of nasolacrimal irrigation at 6 months post-operatively. In patients with tubes these will be removed at 3 months post-operatively. The operation will be considered successful if there is free flow on irrigation with no reflux. It will be considered partially successful if the nasolacrimal duct is patent but there is more than 50% reflux as assessed by an experienced oculoplastic surgeon. It will be considered a failure if there is more than 50% reflux.

The secondary end point will be anatomical success, as measured by patency of nasolacrimal irrigation at 6 months post-operatively.

Statistical analysis planned From a previous study by the PI[1] (and also from numerous other studies in the ophthalmic literature) the baseline success rate for endonasal DCR with tubes is 90%. The current trial is a non-inferiority study, ie to demonstrate that surgery without tubes is not inferior to surgery with tubes.

In order to demonstrate non-inferiority, the recommended approach is to pre-specify a margin of non-inferiority in the protocol. After study completion, a two-sided 95% confidence interval for the true difference between the two agents will be constructed.[8]

Planned sample size A sample size of 200 (100 participants in each arm of the trial) is expected to give a 95% confidence interval of width of approximately 0.15 ie +/- 7.5% around the estimated difference in success rates.

References

1. Dolman PJ. Comparison of external dacryocystorhinostomy with nonlaser endonasal dacryocystorhinostomy. Ophthalmology. 2003 Jan;110(1):78-84
2. Smirnov G, Tuomilehto H, Teräsvirta M, Nuutinen J, Seppä J. Silicone tubing after endoscopic dacryocystorhinostomy: is it necessary? Am J Rhinol. 2006 Nov-Dec;20(6):600-2
3. Mortimore S, Banhegy GY, Lancaster JL, Karkanevatos A. Endoscopic dacryocystorhinostomy without silicone stenting. J R Coll Surg Edinb. 1999 Dec;44(6):371-3
4. Kashkouli MB, Parvaresh M, Modarreszadeh M, Hashemi M, Beigi B. Factors affecting the success of external dacryocystorhinostomy. Orbit. 2003 Dec;22(4):247-55
5. Beigi B, Westlake W, Chang B, Marsh C, Jacob J, Chatfield J. Dacryocystorhinostomy in south west England. Eye. 1998;12 ( Pt 3a):358-62.
6. Unlü HH, Oztürk F, Mutlu C, Ilker SS, Tarhan S. Endoscopic dacryocystorhinostomy without stents. Auris Nasus Larynx. 2000 Jan;27(1):65-71
7. Smirnov G, Tuomilehto H, Teräsvirta M, Nuutinen J, Seppä J. Silicone tubing is not necessary after primary endoscopic dacryocystorhinostomy: A prospective randomized study. Am J Rhinol 22, 214-217, 2008
8. http://www.emea.europa.eu/pdfs/human/ewp/215899en.pdf

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 16 years) undergoing primary DCR for NLDO who have given fully informed consent to be in the trial

Exclusion Criteria:

* Age less than 16 years
* Previous ipsilateral DCR or nasal surgery
* Canalicular disease

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-11; Primary Completion 2016-06-02 (Actual); Study Completion 2016-06-02 (Actual)

PRIMARY OUTCOMES:
The primary end point will be functional success, determined by patient-reported symptoms. This will be assessed a minimum of six months post-operatively. In patients with tubes these will be removed at 3 months post-operatively. | 6 months

SECONDARY OUTCOMES:
The secondary end point will be anatomical success, as measured by patency of nasolacrimal irrigation at 6 months post-operatively. In patients with tubes these will be removed at 3 months post-operatively. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Dolman, MD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - Eye Care Centre (Clinic), Vancouver, British Columbia
  - VGH/UBC (Operating Rooms), Vancouver, British Columbia